CLINICAL TRIAL: NCT03109938
Title: Comparison of Diagnostic Accuracies of Various Endoscopic Examination Techniques for Evaluating the Invasion Depth of Lateral Spreading Tumours (LST).
Brief Title: Comparison of Diagnostic Accuracies of Various Endoscopic Examination Techniques
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: LST2016
Record Dates: First submitted 2017-03-28; First posted 2017-04-12 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endoscopic diagnosis of lateral spreading tumours (LST) with submucosal invasion is important in guiding the treatment strategy. The use of advanced imaging is not standard clinical practice in China. A clinical trial is now under way comparing the accuracy of narrow band imaging (NBI), endoscopic ultrasonography (EUS) and magnifying chromoendoscopy (MCE) for the diagnosis of LST with submucosal invasion.

DETAILED DESCRIPTION:
Endoscopic diagnosis of lateral spreading tumours (LST) with submucosal invasion is important in guiding the treatment strategy. The use of advanced imaging is not standard clinical practice in China. A clinical trial is now under way comparing the accuracy of narrow band imaging (NBI), endoscopic ultrasonography (EUS) and magnifying chromoendoscopy (MCE) for the diagnosis of LST with submucosal invasion.The final histologic diagnosis was used as the true diagnosis in the present study. By comparing the consistency of histologic diagnosis and preoperative evaluation,the diagnostic accuracies of various endoscopic examination techniques(narrow band imaging , endoscopic ultrasonography , and magnifying chromoendoscopy) was calculated respectively.

ELIGIBILITY:
Inclusion Criteria:

- patients older than 18 years and Less than 65 years patients with endoscopic diagnosis of lateral spreading tumours signed informed consent

Exclusion Criteria:

- patients with serious heart, brain, lung, kidney complications patients with intestinal obstruction previous therapy for colorectal cancer women in gestational and lactational period taking anticoagulants or antiplatelet medications. based on the evaluations of physicians, the patient's condition is not suitable for the clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with endoscopic diagnosis of lateral spreading tumours
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracies | one week
  The final histologic diagnosis was used as the true diagnosis in the present study. By comparing the consistency of histologic diagnosis and preoperative evaluation,the diagnostic accuracies of various endoscopic examination techniques(narrow band imaging , endoscopic ultrasonography , and magnifying chromoendoscopy) was calculated respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Baoping Wu, Principal Investigator — Guangdong Provincial Key Laboratory of Gastroenterology
Locations (1):
- Guangdong Provincial Key Laboratory of Gastroenterology,Department of Gastroenterology, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No